CLINICAL TRIAL: NCT06074900
Title: The WHERE Study: Waiting for Hip and KneE REplacement - A Prospective Cohort
Brief Title: The WHERE Study: Waiting for Hip and KneE REplacement
Acronym: WHERE
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 119349
Record Dates: First submitted 2021-10-18; First posted 2023-10-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: TJR; Hip; Knee; Osteoarthiritis; Wait times; Total hip replacement; Total knee replacement
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Prospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: prospective cohort study — This study is observational in nature and does not involve any experimental treatments or additional radiographs, diagnostic tests or clinical interventions beyond what is regularly prescribed within the context of standard of care for each patient.
  Outcomes for participants will be measured and captured primarily during regularly scheduled clinic/hospital visits, which include standard of care clinical examinations. Participants will be asked to complete study questionnaires as per the visit schedule and participant data will be recorded on applicable study CRFs at the appropriate time points. CRFs detailing patient, injury, and treatment variables of interested will be collected at the time of recruitment.

SUMMARY:
Total hip and knee replacements (TJR) for osteoarthritis are common orthopaedic procedures performed in Canada. Waits for these procedures are already common and lengthy, and the COVID-19 pandemic has resulted in the further of delay of thousands of scheduled TJRs. Longer wait times for TJR can be associated with increased pain and functional disability, and up to 80% of patients awaiting TJR use opioids for pain management. Further, pre-operative pain, functional disability and opioid use has been linked to worse recovery and continued opioid abuse post-operatively. Interestingly, some clinical studies have shown that not all patients experience a deterioration in symptoms while on the waitlist for TJR, and a longer wait time is not always associated with poor post-operative outcomes. However, there is insufficient evidence surrounding the relationships between wait time, patient characteristics, and outcomes both prior to and following hip or knee replacement.

The Investigators aim to establish a large prospective cohort of patients with osteoarthritis waiting for TJR with key research questions and the overarching objectives of identifying which patients deteriorate while on the waitlist, and how wait time affects patient-important outcomes following surgery.

The study will enroll 3008 patients awaiting TJR at 10 Centres from across Canada. All participating site investigators are fellowship trained Orthopaedic surgeons, working in acute care facilities with active research programs and dedicated research staff. The study will follow the patients from their waitlist enrolment up to two years post-operatively. During this time, the research team will collect pain, function, opioid use, and quality of life measures at regular intervals. In addition, an economic analysis will be conducted to determine the impact of length of time on a waitlist on patient and healthcare system costs. The data will highlight the consequences of long waits for patients undergoing TJR, information that will improve patient care and provide insight for refining wait list policies.

DETAILED DESCRIPTION:
Understanding the association between sex, gender, SED (socioeconomic deprivation) PD (psychological distress), and the use of NSIs (non- surgical interventions) with distinct trajectories of deterioration prior to TJR, and the interactions between these variables, wait time, and post-operative recovery could help identify patient groups with the greatest unmet needs, and develop appropriate care plans. Effective waitlist management requires tracking the flow of patients as they progress toward surgery to identify patients at high or low risk of deterioration. Identifying those who require enhanced support while awaiting TJR, as well as delineating the relationship between wait time and post-operative outcomes within trajectory subgroups will enable targeted, patient-centered care. Managing waitlists for TJR based on evidence-based, clinically informative subgroups could eliminate inefficiencies and inequities in decision making and smooth the flow of patients. For these reasons, we aim to establish WHERE, the first prospective longitudinal study of patients awaiting TJR with the overarching objective of identifying which patients are most affected by longer waits, and how inequities affect the progression of symptoms prior-to, and recovery following TJR.

Managing waitlists for TJR based on evidence-based, clinically informative subgroups could eliminate inefficiencies and inconsistencies in decision making and smooth the flow of patients. For these reasons, the Investigators aim to establish WHERE, the first prospective cohort study of patients awaiting TJR with targeted research questions, and the overarching objective of identifying which patients deteriorate while on the waitlist and which patients may tolerate longer wait times.

WHERE will be the first prospective study to investigate distinct group-based trajectories of pre-operative pain, functional ability, opioid use, and health resource utilization (HRU) and their association with TJR patient characteristics and post-operative recovery and outcomes. The data collected will outline complex associations between delivery of care and symptoms in a representative setting, identify where performance improvement efforts need to be targeted, allow better identification and treatment of high-risk subgroups, and help set the foundation for creating improved, risk-stratified care pathways.

We have identified the following research questions as priorities to address with the WHERE cohort:

1. What factors are associated with different trajectories of preoperative symptoms and opioid use in patients awaiting TJR?

   There is a paucity of evidence surrounding the trajectory of pre-operative symptoms and functional ability in patients with end-stage OA awaiting TJR, and how these may differ by SED or psychological variables.

   Study Aims:

   i) Determine whether previously identified trajectories of OA symptom progression are reproducible in patients scheduled for TJR in Canada; ii) Describe the relationships between SED and psychological variables with trajectory membership; iii) Identify time points in each sub-group where trajectories significantly change.
2. Could targeted NSIs improve symptom management for patients waiting for TJR? Some patients awaiting TJR may not experience a significant deterioration in symptoms, and as many as 50% of patients undergoing TJR may not be appropriate surgical candidates, suggesting they could benefit from further NSIs prior to being scheduled for TJR.

   Study Aims:

   i) Characterize variation in the use of NSIs prior to TJR; ii) Identify which NSI types alleviate symptoms while awaiting TJR to inform symptom management programs; iii) Determine whether sex, gender, SED, or PD are associated with the use of, barriers to, and satisfaction with NSIs.
3. Is the association between wait time and postoperative outcomes modified by trajectory group? Differences in the progression of symptoms while awaiting TJR may contribute to the inconsistent evidence surrounding the relationship between wait time and postoperative outcomes.

   Study Aims:

   i) Determine how longer wait times impact post-TJR outcomes in different trajectory groups; ii) Identify wait time thresholds within sub-groups to establish evidence-based targets.
4. Does variation in symptom progression, functional deterioration, and opioid use while on the waitlist affect the cost-effectiveness of TJR? No studies have evaluated the cost-effectiveness of TJR for patients with different trajectories of pre-operative pain, functional ability, and opioid use, or the cost-effectiveness of TJR using evidence-based, patient-centered wait time cut-offs.

Study Aims:

i) Provide insight into the association between variable pre-operative symptom trajectories and health-care system costs; ii) Examine the association between patient-centered wait time thresholds within trajectory sub-groups and health-care system costs following TJR.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older;
2. Primary OA of the hip or knee (as defined by the American College of Rheumatology)60,61;
3. Provision of informed consent

Exclusion Criteria:

1. Hip or knee arthritis other than OA;
2. Previous TJR or retained hardware on the ipsilateral side;
3. Refusal to participate;
4. Inability to provide informed consent;
5. Likely to have problems maintaining follow-up in the opinion of the investigator (i.e. no fixed address, severe mental disorders or additions without adequate support
6. Inability to speak or understand English without a registered interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with hip or knee OA booked for a surgical consult at the participating sites will be eligible for inclusion based on the above inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 3008 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported pain and functional ability | 24 months
  Patient-reported pain and functional ability, measured by the Hip/Knee Disability and Osteoarthritis, Joint Replacement scores (H/KOOS-JR).The H/KOOS-JR scores were developed specifically for patients with OA undergoing TJR, and have sufficient measurement properties in OA patients undergoing TJR when administered in person or via telephone.

SECONDARY OUTCOMES:
Prescription opioid use | 24 months
  Measured via the Narcotics Monitoring System
Perceived disability | 24 months
  Measured via the Pain Disability Questionnaire.
Social support | 24 months
  Measured via the modified Medical Outcomes Study-Social Support Scale (MOS-SSS).
Health-related quality of life (HRQOL) | 24 months
  Measured using the patient-reported EuroQol-5D-5L (EQ5D) score.
Physical Activity | 24 months
  Measured via the International Physical Activity Questionnaire short form.
Health Services Utilization (HSU) and costs | 24 months
  Measured using the patient-reported Ambulatory and Home Care Record (AHCR), which assesses the total cost of illness from a societal perspective, and has very high agreement with administrative HSU. In addition, we will obtain administrative HSU and cost data from the databases at the Institute for Clinical Evaluative Sciences (ICES). Costs will include all costs incurred to the Ministry of Health and Long-Term Care (MoHLTC).
Behavioral Pain | 12 and 24 months
  Collected via the Chronic Pain Behavioral Pain Scale (CPBPs), an objective pain scale developed to mitigate over-exaggeration in self-reported pain
Patient global assessment of health | 12 and 24 months
  Collected via a validated Visual Analog Scale (0 = very poor health).
Patient Satisfaction | 12 and 24 months
  Via a valid and reliable patient-reported measure that evaluates patients' satisfaction with their TJR. This measure considers pain relief, ability to do house/yard work or recreational activities, as well as overall satisfaction and how TJR improved their quality of life.
Clinical outcomes (Radiographic and Performance). | 12 and 24 months
  Measured and recorded by a trained, independent assessor where possible, including:
  * Radiographic: Radiolucencies, wear and osteolysis, component loosening, instability, or heterotopic ossification.
  * Performance: The OMERACT-OARSI recommended timed up and go test (TUG), which valid and reliable for patients with hip and knee OA
Complications | As needed.
  Including those detected radiographically (listed above), infection, leg length discrepancy, instability and dislocation, peri-prosthetic fracture, or any re-operations.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No